CLINICAL TRIAL: NCT03115957
Title: Early Versus Delayed Parenteral Nutrition in Abdominal Surgical Patients With Nutritional Risk and Initial Enteral Nutrition Intolerance: A Clinical Randomized Trial
Brief Title: Early Versus Delayed Parenteral Nutrition in Abdominal Surgical Patients
Acronym: PNASIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jinling Hospital, China (Other)
Collaborators: Peking Union Medical College Hospital (Other); Chinese PLA General Hospital (Other); First Affiliated Hospital, Sun Yat-Sen University (Other); Xijing Hospital (Other); West China Hospital (Other); Xinqiao Hospital of Chongqing (Other); Second Affiliated Hospital, School of Medicine, Zhejiang University (Other); Changhai Hospital (Other); Shanghai 10th People's Hospital (Other); The Second Affiliated Hospital of Harbin Medical University (Other); The Affiliated Hospital of Qingdao University (Other); First Affiliated Hospital of Kunming Medical University (Other)
Responsible Party: Principal Investigator, Wang Xinying, Professor, Chief of Clinical Nutrition Service, Jinling Hospital, China
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201502022-22
Record Dates: First submitted 2017-03-30; First posted 2017-04-14 (Actual); Last update posted 2020-09-29 (Actual); Status verified 2020-09

CONDITIONS: Digestive System Neoplasms
Keywords: Parenteral Nutrition; Digestive System Neoplasms; Randomized Controlled Trials; Clinical Outcomes; Postoperative Period
MeSH Terms: conditions — Digestive System Neoplasms; Hyperphagia | interventions — Parenteral Nutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Early PN (Experimental): Patients who can not tolerate 30% of target energy EN will receive supplemental parenteral nutrition at day 3 after abdominal surgery.
  Interventions: Other: Parenteral Nutrition
- Delayed PN (Experimental): Patients who can not tolerate 30% of target energy EN will receive supplemental parenteral nutrition at day 8 after abdominal surgery.
  Interventions: Other: Parenteral Nutrition

INTERVENTIONS:
Other: Parenteral Nutrition — Patients who can not tolerate 30% of target energy EN will receive supplemental parenteral nutrition at day 3 or at day 8 after abdominal surgery.

SUMMARY:
Patients will be randomized to early PN group or late PN group at day 3 after abdominal surgery. Patients will receive supplemental parenteral nutrition or not within 7 days after abdominal surgery. Both groups will receive SPN except 80% of target energy delivered by EN or oral or patients are discharged from hospital. The primary and secondary outcomes will be collected.

DETAILED DESCRIPTION:
Patients after abdominal surgery will attempt enteral nutrition support for 2 days, if she/he can not tolerate 30% of target energy, then she/he will be randomized to early PN group or late PN group at day 3. Patients in early PN group will receive supplemental parenteral nutrition at day 3 while patients in late PN group will not receive supplemental parenteral nutrition until day 8 after abdominal surgery. Both groups will receive SPN except 80% of target energy delivered by EN or oral or patients are discharged from hospital. The primary and secondary outcomes will be collected.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent of patients or their legal representatives to participate in this study.
2. Patients undergoing selective operation without trauma
3. Patients following medium or major abdominal surgery
4. NRS 2002≥ 3

Exclusion Criteria:

1. Psychiatric disorders
2. Pregnancy or breast-feeding women
3. Malnutrition

   1. Weight loss >10%-15% in 6 months
   2. BMI<18.5
   3. SGA score with stage C
   4. Albumin <30g/L
4. Unstable vital signs or unstable hemodynamics (such as systolic blood pressure < 90 mmHg or mean arterial pressure < 70 mmHg after rapid 500 ml crystal or 200 ml gel infusion, or the 50% increase of vascular active drug infusion rate in an hour, etc)
5. Refuse to participate in the study
6. Mortality rates expected to more than 50% in 6 months with malignant or irreversibility diseases

   1. Cancer in terminal stage
   2. HIV positive at end-stage or CD4 < 50/mm3
   3. Cardiopulmonary resuscitation (CPR) before cardiac arrest and nervous system function not fully recovery
   4. Four levels of physical activity of the patients defined by New York heart association
   5. Rely on breathing machine because of chronic diseases
7. Life expectancy less than 24 hours of dying patients
8. Refractory shock to meet any of the following article

   1. The infusion rate of dopamine > 15 ug/kg/min
   2. The infusion rate of dobutamine > 15 ug/kg/min
   3. The infusion rate of epinephrine and norepinephrine > 30 ug/min
   4. The infusion rate of phenylephrine > 50 ug/min
   5. The infusion rate of milrinone > 0.5 ug/kg/min
   6. The infusion rate of vasopressin > 0.04 U/min
   7. Inter aortic ballon pump (IABP)
9. Hepatic insufficiency (alanine/aspartate transaminase 200% above normal range)
10. Renal insufficiency(creatinine 200% above normal range)
11. Metabolic diseases（hyperthyroidism/ hypothyroidism, adrenal cortex disorders)
12. EN can reach 30% of target energy in 48 hours after surgery
13. Burn area exceeding 20% of the patient's body surface
14. Autoimmune diseases or immune dysfunction or history of organ transplantation
15. International standardization ratio (INR) more than 3.0 or platelet count < 30000 cells/mm3 or other hemorrhagic diathesis
16. Intracranial hemorrhage one month before enrolment
17. General contraindications to infusion therapy or history of severe allergy against ingredients of enteral and parenteral nutrition
18. Has already participated in another clinical trial
19. Has started to nutritional support therapy before enrolment
20. Diabetes mellitus (anamnestic and/or under medical treatment)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Actual)
Dates: Start 2017-04-14 (Actual); Primary Completion 2018-12-30 (Actual); Study Completion 2019-02-22 (Actual)

PRIMARY OUTCOMES:
Morbidity of infection | From date of randomization until the date of infection from any cause, assessed up to 2 months.
  Invasion of the host organism by microorganisms that can cause pathological conditions or diseases

SECONDARY OUTCOMES:
Length of stay in hospital | From date of operation until the date of patients discharged from hospital, assessed up to 12 months.
  The length of patients stay in hospital after operation
Mortality | From date of randomization until the date of death, assessed up to 2 months after patients discharged from hospital.
  All deaths reported in all enrolled patients.
Scale the frequency of gastrointestinal intolerance | During the intervention, assessed up to 2 months.
  Diarrhea, vomiting, abdominal distention or cramping and abdominal pain
Scale actual calories intake | During the intervention, assessed up to 2 months.
  The total energy patients received during the intervention
Laboratory examination | At the date of patients enrollment and after intervention, assessed up to 2 months.
  Albumin, pre-albumin, transferrin and retinol conjugated protein

CONTACTS AND LOCATIONS:
Overall Officials: Xinying Wang, MD, Principal Investigator — Jinling Hospital, China
Locations (1):
- JinlingH, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bauer P, Charpentier C, Bouchet C, Nace L, Raffy F, Gaconnet N. Parenteral with enteral nutrition in the critically ill. Intensive Care Med. 2000 Jul;26(7):893-900. doi: 10.1007/s001340051278. PMID 10990103
- [Background] Desachy A, Clavel M, Vuagnat A, Normand S, Gissot V, Francois B. Initial efficacy and tolerability of early enteral nutrition with immediate or gradual introduction in intubated patients. Intensive Care Med. 2008 Jun;34(6):1054-9. doi: 10.1007/s00134-007-0983-6. Epub 2008 Jan 22. PMID 18210092
- [Background] Arabi YM, Tamim HM, Dhar GS, Al-Dawood A, Al-Sultan M, Sakkijha MH, Kahoul SH, Brits R. Permissive underfeeding and intensive insulin therapy in critically ill patients: a randomized controlled trial. Am J Clin Nutr. 2011 Mar;93(3):569-77. doi: 10.3945/ajcn.110.005074. Epub 2011 Jan 26. PMID 21270385
- [Background] Casaer MP, Mesotten D, Hermans G, Wouters PJ, Schetz M, Meyfroidt G, Van Cromphaut S, Ingels C, Meersseman P, Muller J, Vlasselaers D, Debaveye Y, Desmet L, Dubois J, Van Assche A, Vanderheyden S, Wilmer A, Van den Berghe G. Early versus late parenteral nutrition in critically ill adults. N Engl J Med. 2011 Aug 11;365(6):506-17. doi: 10.1056/NEJMoa1102662. Epub 2011 Jun 29. PMID 21714640
- [Background] Rice TW, Mogan S, Hays MA, Bernard GR, Jensen GL, Wheeler AP. Randomized trial of initial trophic versus full-energy enteral nutrition in mechanically ventilated patients with acute respiratory failure. Crit Care Med. 2011 May;39(5):967-74. doi: 10.1097/CCM.0b013e31820a905a. PMID 21242788
- [Background] Singer P, Anbar R, Cohen J, Shapiro H, Shalita-Chesner M, Lev S, Grozovski E, Theilla M, Frishman S, Madar Z. The tight calorie control study (TICACOS): a prospective, randomized, controlled pilot study of nutritional support in critically ill patients. Intensive Care Med. 2011 Apr;37(4):601-9. doi: 10.1007/s00134-011-2146-z. Epub 2011 Feb 22. PMID 21340655
- [Background] National Heart, Lung, and Blood Institute Acute Respiratory Distress Syndrome (ARDS) Clinical Trials Network; Rice TW, Wheeler AP, Thompson BT, Steingrub J, Hite RD, Moss M, Morris A, Dong N, Rock P. Initial trophic vs full enteral feeding in patients with acute lung injury: the EDEN randomized trial. JAMA. 2012 Feb 22;307(8):795-803. doi: 10.1001/jama.2012.137. Epub 2012 Feb 5. PMID 22307571
- [Background] Doig GS, Simpson F, Sweetman EA, Finfer SR, Cooper DJ, Heighes PT, Davies AR, O'Leary M, Solano T, Peake S; Early PN Investigators of the ANZICS Clinical Trials Group. Early parenteral nutrition in critically ill patients with short-term relative contraindications to early enteral nutrition: a randomized controlled trial. JAMA. 2013 May 22;309(20):2130-8. doi: 10.1001/jama.2013.5124. PMID 23689848
- [Background] Heidegger CP, Berger MM, Graf S, Zingg W, Darmon P, Costanza MC, Thibault R, Pichard C. Optimisation of energy provision with supplemental parenteral nutrition in critically ill patients: a randomised controlled clinical trial. Lancet. 2013 Feb 2;381(9864):385-93. doi: 10.1016/S0140-6736(12)61351-8. Epub 2012 Dec 3. PMID 23218813
- [Background] Braunschweig CA, Sheean PM, Peterson SJ, Gomez Perez S, Freels S, Lateef O, Gurka D, Fantuzzi G. Intensive nutrition in acute lung injury: a clinical trial (INTACT). JPEN J Parenter Enteral Nutr. 2015 Jan;39(1):13-20. doi: 10.1177/0148607114528541. Epub 2014 Apr 9. PMID 24722769
- [Background] Charles EJ, Petroze RT, Metzger R, Hranjec T, Rosenberger LH, Riccio LM, McLeod MD, Guidry CA, Stukenborg GJ, Swenson BR, Willcutts KF, O'Donnell KB, Sawyer RG. Hypocaloric compared with eucaloric nutritional support and its effect on infection rates in a surgical intensive care unit: a randomized controlled trial. Am J Clin Nutr. 2014 Nov;100(5):1337-43. doi: 10.3945/ajcn.114.088609. Epub 2014 Sep 3. PMID 25332331
- [Background] Peake SL, Davies AR, Deane AM, Lange K, Moran JL, O'Connor SN, Ridley EJ, Williams PJ, Chapman MJ; TARGET investigators and the Australian and New Zealand Intensive Care Society Clinical Trials Group. Use of a concentrated enteral nutrition solution to increase calorie delivery to critically ill patients: a randomized, double-blind, clinical trial. Am J Clin Nutr. 2014 Aug;100(2):616-25. doi: 10.3945/ajcn.114.086322. Epub 2014 Jul 2. PMID 24990423
- [Background] Petros S, Horbach M, Seidel F, Weidhase L. Hypocaloric vs Normocaloric Nutrition in Critically Ill Patients: A Prospective Randomized Pilot Trial. JPEN J Parenter Enteral Nutr. 2016 Feb;40(2):242-9. doi: 10.1177/0148607114528980. Epub 2014 Apr 3. PMID 24699555
- [Derived] Gao X, Zhang Y, Qi X, Xiao Y, Gao T, Jin G, Wang K, Zhou Y, Chi Q, Yang H, Li M, Yu J, Qin H, Tang Y, Wu X, Li G, Zhang L, Wang X. Early enteral nutrition versus early supplemental parenteral nutrition in patients undergoing major abdominal surgery: a secondary analysis of 2 randomized clinical trials. Am J Clin Nutr. 2024 Apr;119(4):1036-1043. doi: 10.1016/j.ajcnut.2024.02.006. Epub 2024 Feb 17. PMID 38369126
- [Derived] Gao X, Zhang L, Zhang Y, Zhou D, Gao T, Liu Y, Jin G, Wang K, Zhou Y, Chi Q, Yang H, Li M, Yu J, Qin H, Tang Y, Wu X, Li G, Wang X. Effect of early achievement of energy target by different nutritional support strategies on nosocomial infections in patients undergoing major abdominal surgery: a secondary analysis of two randomized clinical trials. Int J Surg. 2023 Sep 1;109(9):2680-2688. doi: 10.1097/JS9.0000000000000526. PMID 37300882
- [Derived] Gao X, Liu Y, Zhang L, Zhou D, Tian F, Gao T, Tian H, Hu H, Gong F, Guo D, Zhou J, Gu Y, Lian B, Xue Z, Jia Z, Chen Z, Wang Y, Jin G, Wang K, Zhou Y, Chi Q, Yang H, Li M, Yu J, Qin H, Tang Y, Wu X, Li G, Li N, Li J, Pichard C, Wang X. Effect of Early vs Late Supplemental Parenteral Nutrition in Patients Undergoing Abdominal Surgery: A Randomized Clinical Trial. JAMA Surg. 2022 May 1;157(5):384-393. doi: 10.1001/jamasurg.2022.0269. PMID 35293973